CLINICAL TRIAL: NCT06493383
Title: Lotrafilcon B Plano Cosmetic Contact Lenses Post-Market Clinical Follow-Up Study
Brief Title: Lotrafilcon B Plano Cosmetic Contact Lenses Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Information to be gathered in survey format instead of a clinical investigation.
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLT354-P001
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cosmetic Appearance
Keywords: Eye color; Colored contact lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AIR OPTIX COLORS (Experimental): Lotrafilcon B plano cosmetic contact lenses worn in both eyes at least 5 hours per day, at least 2 days a week, for one year. Lenses will be replaced monthly and cleaned, rinsed, disinfected, and stored in accordance with the package labeling of the lens care products recommended by the eye care professional.
  Interventions: Device: Lotrafilcon B plano cosmetic contact lenses

INTERVENTIONS:
Device: Lotrafilcon B plano cosmetic contact lenses — Commercially approved colored contact lenses worn for cosmetic purposes to alter or enhance the apparent color of the eye

SUMMARY:
The purpose of this study is to gather long-term performance and safety data on AIR OPTIX™ COLORS (lotrafilcon B) plano cosmetic contact lenses in subjects 12 years of age and older. AIR OPTIX™ COLORS plano contact lenses do not contain visual correction and are worn for cosmetic purposes only.

DETAILED DESCRIPTION:
Eligible participants will receive the contact lens color of their choice (if available) to be used as intended by the manufacturer for the duration of their participation in the study, approximately 1 year.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject and/or parents/legally authorized representative must be able to understand and sign an approved informed consent form.
* Has never worn contact lenses before, with or without refractive error correction.
* Willing to wear cosmetic contact lenses and who have expressed interest in 1 to 3 color variants of lotrafilcon B plano cosmetic contact lenses.
* Willing to wear the study lenses at least 5 hours per day for at least 2 days a week during the study.
* Best Corrected Visual Acuity (BCVA) of 20/25 or better in each eye at screening.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Any ocular disease or condition that would contraindicate contact lens wear.
* Pregnant and lactating women.
* Any use of systemic or ocular medications that would contraindicate contact lens wear.
* Other protocol-defined exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of corneal infiltrative events | Up to Year 1
  A corneal infiltrate is a single or group of inflammatory cells in the normally clear cornea.
Incidence of microbial keratitis | Up to Year 1
  Microbial keratitis is a sight-threatening infection of the cornea.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No